CLINICAL TRIAL: NCT06428110
Title: Personalized Medication Research of Warfarin Based on Vascular Aging Assessment
Brief Title: A Prospective Cohort Study on Warfarin Personalized Medication
Status: Completed | Type: Observational
Sponsor: Haobin Li (Other)
Responsible Party: Sponsor-Investigator, Haobin Li, Principal Investigator, Shanghai 5th People's Hospital
Organization: Shanghai 5th People's Hospital (Other)
Other Study IDs: 2020081
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Warfarin Sodium Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients taking warfarin with vascular aging group
- Patients taking warfarin with normal vascular group

INTERVENTIONS:
Other:

SUMMARY:
Analyze the impact of the degree of blood vessel aging on the anticoagulant effect and bleeding risk of warfarin. Evaluating the possibility of using the degree of blood vessel aging to guide individualized use of the anticoagulant drug warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older, taking warfarin, with or without premature vascular aging, regardless of gender.

  * Patients who have not concurrently or intermittently used anticoagulant drugs, including antiplatelet drugs, heparin, low molecular weight heparin, and non-vitamin K-dependent oral anticoagulants, such as dabigatran and apixaban.

    * Signing an informed consent form before blood sample collection.

Exclusion Criteria:

* Patients who are allergic to warfarin or lactose.

  * Patients who are receiving immunosuppressive agents or low molecular weight heparin anticoagulants.

    * Patients with bleeding tendencies, blood disorders with platelet counts > 400 × 10^9 /L or < 100 × 10^9 /L, hemoglobin > 169 or < 100 g/L.

      * History of peptic ulcer disease.

        * Malignant tumors, severe multi-organ dysfunction or failure such as heart, liver, and kidney.

          * Neurological disorders such as epilepsy.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients taking warfarin
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Numbers of patients with bleeding events | 1 year during the follow-up
  Numbers of patients with bleeding events during warfarin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guangchun Sun, Principal Investigator — The Fifth People's Hospital of Shanghai
Locations (1):
- The Fifth People's Hospital of Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No